CLINICAL TRIAL: NCT03392818
Title: An Innovative Approach for Accurately Predicting the Optimal Insertion Depth of Uniblocker Without Fiberoptic Bronchoscope Assistance
Brief Title: An Innovative Approach for Uniblocker Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 966169
Record Dates: First submitted 2017-12-24; First posted 2018-01-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Therapeutic Procedural Complication
MeSH Terms: interventions — Food, Formulated

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- formula (Experimental): Calculate the depth of intubation according to the formula of 0.1977* patient's height - 4.2423
  Interventions: Other: formula
- Fiberoptic bronchoscope (Experimental): intubation of Uniblocker under the Under the guidance of Fiberoptic bronchoscope
  Interventions: Device: Fiberoptic bronchoscope
- The measured distance (Experimental): To measure the distance between the upper edge of the thyroid cartilage to the upper edge of the sternum add the distance from the upper edge of the sternum to the carina calculated according to the chest CT scans as a guide to the placement of Uniblocker without the aid of FOB.
  Interventions: Other: The measured distance

INTERVENTIONS:
Other: The measured distance — To measure the distance between the upper edge of the thyroid cartilage to the upper edge of the sternum add the distance from the upper edge of the sternum to the carina calculated according to the chest CT scans as a guide to the placement of Uniblocker without the aid of Fiberoptic bronchoscope.
  Arms: The measured distance
Other: formula — Calculate the depth of intubation according to the formula of 0.1977* patient's height - 4.2423
  Arms: formula
Device: Fiberoptic bronchoscope — The intubation of Uniblocker under the guidance of Fiberoptic bronchoscope
  Arms: Fiberoptic bronchoscope

SUMMARY:
To measure the distance between the upper edge of the thyroid cartilage to the upper edge of the sternum add the distance from the upper edge of the sternum to the carina was calculated according to the chest CT scans as a guide to the placement of Uniblocker without the aid of FOB.

DETAILED DESCRIPTION:
In previous study, the investigators found Chest computed tomography (CT) image can accurately predicting the optimal insertion depth of Uniblocker,however in some hospital the CT scan performed for the preoperative surgical evaluation without the vocal cords slices. If a more extensive CT scan was needed for obtaining a more reliable image of the vocal cords,the additional exposure dose would be a major disadvantage of the method.So the investigators measure the distance between the upper edge of the thyroid cartilage to the upper edge of the sternum add the distance from the upper edge of the sternum to the carina calculated according to the chest CT scans as a guide to the placement of Uniblocker without the aid of FOB.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients undergoing left side thoracic surgery
2. The thoracic surgery requiring a Uniblocker for one-lung ventilation

Exclusion Criteria:

1. Age>70 or <18 years
2. ASA classifications >III
3. BMI >35kg/m2
4. Modified Mallampati classification ≥III
5. Thoracic surgery within the last one month
6. Severe cardiopulmonary disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-07 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The intubation time | 1 year
  The intubation time defined as the time from the anesthesiologist inserted the video laryngoscope between the teeth of patients until Uniblocker at the optimal position and this was done using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Ximing Qi, Study Director — The First Hospital of Qinhuangdao
Locations (1):
- The first hospital of Qinhuangdao, Qinhuangdao, Hebei, China